CLINICAL TRIAL: NCT07192042
Title: Investigation of Using Non-Wearable Devices to Assess Sleep- Disordered Breathing in Hospitalized Patients With Schizophrenia
Acronym: IUNWD
Status: Recruiting | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202505085
Record Dates: First submitted 2025-08-24; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia and Schizophrenia Spectrum Psychosis
Keywords: Schizophrenia; Sleep- Disordered Breathing; Obstructive Sleep Apnea; Non-Wearable Devices; Hospitalized Patients
MeSH Terms: conditions — Schizophrenia; Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: schizophrenia

SUMMARY:
This research project aims to evaluate the prevalence of comorbid OSA and its impact on disease progression among hospitalized schizophrenia patients using non-wearable devices.

DETAILED DESCRIPTION:
Schizophrenia patients frequently experience sleep disorders and circadian rhythm disruptions, with Obstructive Sleep Apnea (OSA) being particularly prevalent. Evidence indicates that schizophrenia patients have approximately twice the risk of developing OSA compared to the general population, and comorbid OSA may worsen clinical outcomes, reduce quality of life, and increase mortality. Traditional OSA diagnosis relies on overnight Polysomnography (PSG), which is costly, difficult to implement, and associated with lower compliance among psychiatric patients, leading to delayed detection and treatment.

This study aims to evaluate the prevalence of comorbid OSA and its impact on disease progression in hospitalized schizophrenia patients using non-wearable monitoring devices. A smart sensing pad based on Noninvasive Fiber Optic Physiological Monitoring Technology (nFOPT) will be employed to capture sleep physiological signals, while OSA severity will be compared with assessments from a simplified sleep-disordered breathing screening device (Belun Ring). The study will incorporate clinical psychiatric symptom evaluations, nurses' observations recorded every 30 minutes during hospitalization, and data from wearable bands capturing daytime activity levels and sleep behaviors. Statistical and machine learning analyses will be applied to examine correlations between OSA severity and changes in psychiatric symptoms and to develop multimodal prediction models.

Expected outcomes include: (1) determination of the prevalence and severity distribution of OSA among hospitalized schizophrenia patients, (2) characterization of the relationship between OSA severity and psychiatric symptom changes, and (3) validation of non-wearable fiber optic monitoring technology for early screening and risk prediction. The application of clinically feasible, non-wearable devices is intended to enhance detection of comorbid sleep-disordered breathing in schizophrenia and support timely diagnostic and therapeutic interventions, ultimately improving patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 20 and 70 years old.
* Diagnostic Criteria: Schizophrenia spectrum disorders, including schizophrenia, schizoaffective disorder, and schizophreniform disorder, diagnosed according to DSM-5 criteria and confirmed with the MINI 7.0 (Chinese version).
* Clinical Stability and Informed Consent: At the time of admission, participants should be in a relatively stable condition, able to understand the study procedures, and capable of providing written informed consent. If patients are unable to fully comprehend due to illness severity or cognitive limitations, consent may be obtained from a legal guardian or family member, with subsequent confirmation of consent by the patient once their condition improves.

Exclusion Criteria:

* Treatment-related: Patients who are currently receiving continuous positive airway pressure (CPAP) therapy for OSA.
* Other Major Central Nervous System Disorders: Presence of other serious conditions that may significantly affect central nervous system function, aside from schizophrenia, such as major depressive disorder or bipolar disorder.
* Severe Medical Illnesses: Including, but not limited to, malignant tumors, end-stage cardiopulmonary disease, neuromuscular disorders severely affecting motor or respiratory function, uncontrolled epileptic seizures, or other serious medical conditions that prevent patients from sleeping in the supine position.
* Clinical Judgment: Patients deemed unsuitable for participation due to clinical conditions (e.g., agitation, non-cooperation, or other safety concerns).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with schizophrenia in the acute psychiatric ward at Shuang Ho Hospital, TMU, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Exploring the Prevalence of Obstructive Sleep Apnea (OSA) in Patients with Schizophrenia | From Day 1 through study completion, an average of 3 weeks
  The prevalence and distribution of OSA across different severity levels will be evaluated using the apnea-hypopnea index/respiratory event index derived from the Belun Ring (bAHI). Belun Ring is a wearable, non-invasive device designed to continuously monitor physiological signals during daily life and sleep. It uses optical and motion sensors to provide detailed data on autonomic and sleep-related parameters. The severity of OSA is categorized based on the bAHI as follows: Normal: bAHI < 5 events/hour; Mild OSA: bAHI between 5 and 15 events/hour; Moderate OSA: bAHI between 15 and 30 events/hour; Severe OSA: bAHI > 30 events/hour.
Non-invasive Fiber Optic Physiological Monitoring (nFOPT) for respiratory patterns | From Day 1 through study completion, an average of 3 weeks
  A novel non-invasive monitoring technique that uses fiber optic sensors to continuously measure physiological signals with high sensitivity and stability. This technology aims to investigate respiratory patterns during sleep. Higher irregularity in respiratory patterns may indicate poorer physiological regulation, while stable and coherent signals suggest healthier sleep and autonomic function.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | From Day 1 through study completion, an average of 3 weeks
  A clinician-administered scale designed to assess the severity of positive, negative, and general psychopathology symptoms in schizophrenia. The PANSS consists of 30 items rated on a 7-point Likert scale (1 = absent to 7 = extreme). Total scores range from 30 to 210, with higher scores indicating more severe psychiatric symptoms. Subscales include:
  Positive symptom scale (7 items): evaluates hallucinations, delusions, and other positive symptoms.
  Negative symptom scale (7 items): evaluates blunted affect, social withdrawal, and other negative symptoms.
  General psychopathology scale (16 items): evaluates mood, anxiety, cognitive symptoms, and other general psychopathology.
  Higher total or subscale scores indicate greater symptom severity. The PANSS is widely used to monitor symptom changes during hospitalization or intervention.
Brief Psychiatric Rating Scale (BPRS) | From Day 1 through study completion, an average of 3 weeks
  A clinician-administered scale designed to assess psychiatric symptom severity in patients with schizophrenia and other psychotic disorders. The BPRS includes 18-24 items (depending on version), each rated on a 7-point Likert scale (1 = not present to 7 = extremely severe). Key symptom domains include:
  Positive symptoms: hallucinations, delusions, thought disorder. Negative symptoms: emotional withdrawal, blunted affect, motor retardation. Affective symptoms: anxiety, depression, hostility. Total scores range from 18 (minimal symptoms) to 126 (maximum symptom severity), with higher scores indicating greater symptom severity. The BPRS is commonly used to monitor changes in psychiatric symptoms over time and in response to interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol